CLINICAL TRIAL: NCT00049296
Title: Phase I Pharmacokinetic Trial of Thalidomide and Docetaxel: A Regimen Based on Anti-Angiogenic Therapeutic Principles
Brief Title: Thalidomide and Docetaxel in Treating Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Scot C. Remick, MD, Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CWRU4Y01; P30CA043703 (NIH); CWRU-4Y01; NCI-G02-2123
Record Dates: First submitted 2002-11-12; First posted 2003-01-27 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-06

CONDITIONS: Cancer
Keywords: adult anaplastic astrocytoma; male breast cancer; adult anaplastic oligodendroglioma; adult meningeal hemangiopericytoma; adult brain stem glioma; adult central nervous system germ cell tumor; adult choroid plexus tumor; adult craniopharyngioma; adult ependymoblastoma; adult glioblastoma; adult pilocytic astrocytoma; adult anaplastic ependymoma; adult medulloblastoma; adult meningioma; adult pineoblastoma; adult pineocytoma; adult subependymoma; adult myxopapillary ependymoma; advanced adult primary liver cancer; anterior urethral cancer; carcinoma of the appendix; chondrosarcoma; classic Kaposi sarcoma; AIDS-related Kaposi sarcoma; immunosuppressive treatment related Kaposi sarcoma; recurrent Kaposi sarcoma; clear cell sarcoma of the kidney; disseminated neuroblastoma; extensive stage small cell lung cancer; gastrointestinal stromal tumor; metastatic gastrointestinal carcinoid tumor; metastatic osteosarcoma; metastatic transitional cell cancer of the renal pelvis and ureter; metastatic Ewing sarcoma/peripheral primitive neuroectodermal tumor; adult mixed glioma; ovarian sarcoma; posterior urethral cancer; primary central nervous system lymphoma; pulmonary carcinoid tumor; recurrent adenoid cystic carcinoma of the oral cavity; recurrent adult brain tumor; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Burkitt lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult primary liver cancer; recurrent adult soft tissue sarcoma; recurrent anal cancer; recurrent basal cell carcinoma of the lip; recurrent bladder cancer; recurrent breast cancer; recurrent colon cancer; recurrent esophageal cancer; recurrent esthesioneuroblastoma of the paranasal sinus and nasal cavity; recurrent extrahepatic bile duct cancer; recurrent gallbladder cancer; recurrent gastric cancer; recurrent gastrointestinal carcinoid tumor; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent inverted papilloma of the paranasal sinus and nasal cavity; recurrent lymphoepithelioma of the nasopharynx; recurrent lymphoepithelioma of the oropharynx; recurrent mantle cell lymphoma; recurrent melanoma; recurrent metastatic squamous neck cancer with occult primary; recurrent midline lethal granuloma of the paranasal sinus and nasal cavity; recurrent mucoepidermoid carcinoma of the oral cavity; recurrent neuroblastoma; recurrent non-small cell lung cancer; recurrent osteosarcoma; recurrent pancreatic cancer; recurrent rectal cancer; recurrent renal cell cancer; recurrent small cell lung cancer; recurrent small intestine cancer; recurrent squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent transitional cell cancer of the renal pelvis and ureter; recurrent Ewing sarcoma/peripheral primitive neuroectodermal tumor; recurrent urethral cancer; recurrent uterine sarcoma; recurrent verrucous carcinoma of the larynx; recurrent verrucous carcinoma of the oral cavity; refractory multiple myeloma; rhabdoid tumor of the kidney; small intestine adenocarcinoma; small intestine leiomyosarcoma; small intestine lymphoma; stage II esophageal cancer; stage II pancreatic cancer; stage III esophageal cancer; stage III multiple myeloma; stage III pancreatic cancer; stage IV adenoid cystic carcinoma of the oral cavity; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult Burkitt lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV anal cancer; stage IV basal cell carcinoma of the lip; stage IV bladder cancer; stage IV breast cancer; stage IV colon cancer; stage IV esophageal cancer; stage IV esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage IV gastric cancer; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV inverted papilloma of the paranasal sinus and nasal cavity; stage IV lymphoepithelioma of the nasopharynx; stage IV lymphoepithelioma of the oropharynx; stage IV mantle cell lymphoma; stage IV melanoma; stage IV midline lethal granuloma of the paranasal sinus and nasal cavity; stage IV mucoepidermoid carcinoma of the oral cavity; stage IV non-small cell lung cancer; stage IV rectal cancer; stage IV renal cell cancer; stage IV squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV uterine sarcoma; stage IV verrucous carcinoma of the larynx; stage IV verrucous carcinoma of the oral cavity; unresectable extrahepatic bile duct cancer; unresectable gallbladder cancer; unspecified adult solid tumor, protocol specific; urethral cancer associated with invasive bladder cancer; recurrent salivary gland cancer; stage IV salivary gland cancer; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; stage IV adult soft tissue sarcoma; adult grade III meningioma; adult oligodendroglioma; adult giant cell glioblastoma; adult gliosarcoma; stage IV pancreatic cancer
MeSH Terms: conditions — Neoplasms; Astrocytoma; Breast Neoplasms, Male; Oligodendroglioma; Choroid Plexus Neoplasms; Craniopharyngioma; Neuroectodermal Tumors, Primitive; Glioblastoma; Ependymoma; Medulloblastoma; Meningioma; Pinealoma; Glioma, Subependymal; Appendiceal Neoplasms; Chondrosarcoma; AIDS-related Kaposi sarcoma; Sarcoma, Kaposi; Gastrointestinal Stromal Tumors; Osteosarcoma; Neuroectodermal Tumors, Primitive, Peripheral; Glioma; Brain Neoplasms; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Burkitt Lymphoma; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Carcinoma, Hepatocellular; Sarcoma; Anus Neoplasms; Urinary Bladder Neoplasms; Breast Neoplasms; Colonic Neoplasms; Esophageal Neoplasms; Esthesioneuroblastoma, Olfactory; Bile Duct Neoplasms; Gallbladder Neoplasms; Stomach Neoplasms; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Melanoma; Neuroblastoma; Carcinoma, Non-Small-Cell Lung; Pancreatic Neoplasms; Rectal Neoplasms; Carcinoma, Renal Cell; Small Cell Lung Carcinoma; Squamous Cell Carcinoma of Head and Neck; Urethral Neoplasms; Multiple Myeloma; Salivary Gland Neoplasms; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Gliosarcoma | interventions — Docetaxel; Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: docetaxel — Patients receive docetaxel IV over 30 minutes once weekly. Courses repeat every 12 weeks in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of docetaxel and thalidomide until the maximum tolerated dose (MTD) is determined.
Drug: thalidomide — Patients receive oral thalidomide twice daily. Courses repeat every 12 weeks in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of docetaxel and thalidomide until the maximum tolerated dose (MTD) is determined.
  Other Names: alpha-phthalimidoglutarimide; N-phthaloylglutamimide; N-phthalylglutamic acid imide

SUMMARY:
RATIONALE: Thalidomide may stop the growth of cancer by stopping blood flow to the tumor. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining thalidomide with docetaxel may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combining thalidomide with docetaxel in treating patients who have advanced cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of docetaxel when administered with thalidomide in patients with advanced solid tumors, multiple myeloma, and non-Hodgkin's lymphoma.
* Determine the dose-limiting toxicity and safety profile of this regimen in these patients.
* Determine the plasma pharmacokinetics of this regimen in these patients.
* Determine the objective tumor response and prolonged freedom from progression in patients treated with this regimen.

OUTLINE: This is a dose-escalation study.

Patients receive oral thalidomide twice daily and docetaxel IV over 30 minutes once weekly. Courses repeat every 12 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of docetaxel and thalidomide until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 1 of 3 or 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: A total of 3-30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignancy not amenable to curative surgery, radiotherapy, or chemotherapy
* Tumor types may include any of the following:

  * Any solid tumor including, but not limited to, head and neck, breast, lung, gastrointestinal, genitourinary, melanoma, and sarcoma
  * Primary CNS neoplasms if the following are true:

    * Received primary radiotherapy
    * No concurrent corticosteroids or has been on a stable corticosteroid dose for at least 30 days
    * No concurrent enzyme-inducible anti-epileptic medications (i.e., carbamazepine or phenytoin)
  * Multiple myeloma
  * Non-Hodgkin's lymphoma
* No refractory or relapsed acute or chronic leukemia
* Measurable or evaluable disease
* No life-prolonging therapy available
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Male or female

Menopausal status

* Not specified

Performance status

* ECOG 0-1

Life expectancy

* At least 4 months

Hematopoietic

* WBC at least 4,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic

* Bilirubin no greater than upper limit of normal (ULN)
* AST and/or ALT no greater than 2.5 times ULN if alkaline phosphatase less than ULN OR
* Alkaline phosphatase no greater than 4 times ULN if AST/ALT less than ULN

Renal

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance at least 60 mL/min

Cardiovascular

* No New York Heart Association class III or IV heart disease

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 2 effective methods of contraception 4 weeks before, during, and 4 weeks after study
* Willing and able to comply with FDA-mandated STEPS program
* No peripheral neuropathy grade 2 or greater
* No prior severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* No more than 2 prior courses of mitomycin

Endocrine therapy

* See Disease Characteristics

Radiotherapy

* At least 4 weeks since prior large-field radiotherapy and recovered

Surgery

* Not specified

Other

* At least 3 weeks since other prior anticancer therapy and recovered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2002-07; Primary Completion 2004-12 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose of docetaxel when administered with thalidomide in patients with advanced solid tumors, multiple myeloma, and non-Hodgkin's lymphoma. | Weekly courses repeat every 12 weeks in the absence of disease progression or unacceptable toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Scot C. Remick, MD, Principal Investigator — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Locations (1):
- Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

REFERENCES:
- [Result] Sanborn SL, Cooney MM, Dowlati A, Brell JM, Krishnamurthi S, Gibbons J, Bokar JA, Nock C, Ness A, Remick SC. Phase I trial of docetaxel and thalidomide: a regimen based on metronomic therapeutic principles. Invest New Drugs. 2008 Aug;26(4):355-62. doi: 10.1007/s10637-008-9137-0. Epub 2008 May 10. PMID 18470481